CLINICAL TRIAL: NCT04043520
Title: Bioenergetic and Metabolic Consequences of the Loss of Ovarian Function in Women - 2018
Brief Title: Bioenergetic Effects of Aging and Menopause (BEAM)
Acronym: BEAM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 18-2483; U54AG062319 (NIH)
Record Dates: First submitted 2019-06-25; First posted 2019-08-02 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Menopause; Obesity, Abdominal; Aging; Weight Gain
MeSH Terms: conditions — Obesity, Abdominal; Weight Gain | interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Postmenopausal: GnRH antagonist + estradiol (Experimental): GnRH antagonist is degarelix acetate, 80 mg, delivered twice as a subcutaneous injection (at baseline and after 12 weeks)
  Estradiol is a transdermal patch 0.075 mg, applied weekly for 24 weeks
  Interventions: Drug: GnRH antagonist; Drug: Estrogen Product
- Postmenopausal: GnRH antagonist + placebo (Experimental): GnRH antagonist is degarelix acetate, 80 mg, delivered twice as a subcutaneous injection (at baseline and after 12 weeks)
  Placebo is a transdermal patch, applied weekly for 24 weeks
  Interventions: Drug: GnRH antagonist; Drug: Placebo estradiol
- Postmenopausal: placebo + placebo (Placebo Comparator): Placebo (1) is normal saline, delivered twice as a subcutaneous injection (at baseline and after 12 weeks)
  Placebo (2) is a transdermal patch, applied weekly for 24 weeks
  Interventions: Drug: Placebo estradiol; Drug: Placebo GnRH antagonist

INTERVENTIONS:
Drug: GnRH antagonist — GnRH antagonist will be given once for premenopausal women (12-week intervention) and twice for postmenopausal women (24-week intervention)
  Other Names: Degarelix Acetate
  Arms: Postmenopausal: GnRH antagonist + estradiol; Postmenopausal: GnRH antagonist + placebo
Drug: Estrogen Product — Estrogen patches will be worn by those randomized to the Estradiol arms in both premenopausal and postmenopausal groups. Patches will be applied weekly and will be worn for the for entirety of the intervention (12 or 24 weeks).
  Other Names: Estrogen transdermal patch
  Arms: Postmenopausal: GnRH antagonist + estradiol
Drug: Placebo estradiol — Placebo patches will be worn by those randomized to the placebo arms in both premenopausal and postmenopausal groups. Patches will be applied weekly and will be worn for the for entirety of the intervention (12 or 24 weeks).
  Other Names: Placebo transdermal patch
  Arms: Postmenopausal: GnRH antagonist + placebo; Postmenopausal: placebo + placebo
Drug: Placebo GnRH antagonist — Postmenopausal women randomized to the placebo injection arm will receive two placebo drug injections of normal saline (24-week intervention)
  Other Names: Placebo injection
  Arms: Postmenopausal: placebo + placebo

SUMMARY:
The menopause transition is associated with increased risk for weight gain and a shift toward storing fat in the belly region, which may increase risk for cardiovascular disease and diabetes. The study will determine whether the stress hormone cortisol contributes to this shift.

DETAILED DESCRIPTION:
The menopause transition is associated with increased risk for weight gain and a shift toward storing fat in the belly region, which may increase risk for cardiovascular disease and diabetes. The stress hormone cortisol is known to promote the accumulation of belly fat, and there is evidence that low estrogen is associated with higher cortisol levels. The first aim of the study is to determine whether low estrogen levels in premenopausal and early postmenopausal women increase cortisol levels in the blood and in fat tissue. When estrogen level decreases at the time of menopause, there is an increase in follicle-stimulating hormone, or FSH. Recent evidence in mice suggests that blocking FSH prevents the increase in belly fat. The second aim of the study is to determine whether decreasing the high FSH level in postmenopausal women causes a decrease in belly fat and changes other factors that are typically thought to be related to estrogen rather than FSH. Because estrogen and FSH levels fluctuate in premenopausal and early postmenopausal women, the investigators will use an approach that controls estrogen and FSH levels to address the aims. The investigators will use a drug that is typically used to treat endometriosis or uterine fibroids to reduce estrogen and FSH levels and an estrogen patch to increase estrogen in some women. The study will generate new knowledge on how menopause affects fat gain and disease risk.

ELIGIBILITY:
Inclusion Criteria:

Volunteers will be healthy peri/postmenopausal women who are willing and able to undergo the proposed hormone manipulation and study procedures. Women will be at least 6 months but not more than 7 years past the last menstrual period (i.e., late perimenopausal or early postmenopausal) with FSH >30 IU/L. We will make a major effort to ensure that the women enrolled in this study come from all races and ethnicities and a wide range of socioeconomic and educational levels. Women will be excluded for the reasons listed below.

Exclusion Criteria:

* abnormal vaginal bleeding
* on hormonal contraceptive or menopausal therapy or intention to start during the period of study
* positive pregnancy test or intention to become pregnant during the period of study
* lactation
* known hypersensitivity to degarelix acetate, estradiol, or medroxyprogesterone acetate
* Center for Epidemiological Studies Depression Scale (CES-D) score <,16 (unless clinician follow-up and clinical judgement determine they are eligible (will be noted in study chart)
* current tobacco and/or vape use more than 2 times/week
* current marijuana or tetrahydrocannabinol (THC) use in any form more than 3 times/week
* regular self-reported alcohol consumption >14 drinks/week
* BMI >39 kg/m2
* use of glucocorticoids or drugs that affect glucocorticoid metabolism (e.g., ketoconazole)
* severe osteopenia or osteoporosis, defined as femoral neck or lumbar spine t-score <-2.0
* thyroid dysfunction, defined as an ultrasensitive TSH <0.5 or >5.0 mU/L; volunteers with abnormal thyroid stimulating hormone (TSH) values will be re-considered for participation in the study after follow-up evaluation by the PCP with initiation or adjustment of thyroid hormone replacement
* liver dysfunction, defined as liver function tests (AST, ALT) >1.5 times the upper limit of normal
* uncontrolled hypertension defined as resting systolic BP >150 mmHg or diastolic BP>90 mmHg; participants who do not meet these criteria at first screening will be re-evaluated, including after follow-up evaluation by the primary care provider (PCP) with initiation or adjustment of anti-hypertensive medications
* self-reported history of breast cancer or other estrogen-dependent neoplasms
* self-reported history of venous thromboembolism, pulmonary embolism, or other thromboembolic disorder
* self-reported history of cardiovascular disease

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2019-09-24 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in the Microdialysis Cortisone Challenge (MCC) Index | Baseline, week 12
  The MCC Index is an in vivo measurement of local cortisol production in abdominal adipose tissue. A higher MCC Index is an indicator of more local cortisol production.
Change in the Oral Cortisone Challenge (OCC) Area Under the Curve (AUC) | Baseline, week 12
  The OCC AUC is a systemic measurement of peripheral glucocorticoid metabolism. A higher OCC AUC is an indicator of more production of cortisol.

SECONDARY OUTCOMES:
Change in lumbar spine Bone Mineral Density (BMD) | Baseline, week 24
  Lumbar spine BMD is measured by dual-energy x-ray absorptiometry. A higher BMD is a general indicator of less risk for osteoporosis.
Change in resting energy expenditure (REE) | Baseline, week 12, week 24
  REE is an index of metabolic rate at rest, measured by indirect calorimetry. A higher REE is an indicator of greater energy expenditure at rest.
Change in visceral fat area (VFA) | Baseline, week 24
  VFA of the abdominal visceral region is measured by computed tomography. VFA is an indicator of the amount of fat stored in this region.
Change in flow-mediated dilation (FMD) | Baseline, week 12, week 24
  FMD of the brachial artery as an index of vascular function. A higher number is a general indicator of better vascular function.
Change in proximal femur Bone Mineral Density (BMD) | Baseline, week 24
  Proximal femur BMD is measured by dual-energy x-ray absorptiometry. A higher BMD is a general indicator of less risk for osteoporosis.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy M Kohrt, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado - Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No